CLINICAL TRIAL: NCT03911128
Title: A Treatment Study Protocol of the ALLTogether Consortium for Infants, Children and Young Adults (0-45 Years of Age) With Newly Diagnosed Acute Lymphoblastic Leukaemia (ALL): a Pilot Study
Brief Title: A Treatment Protocol for Participants 0-45 Years With Acute Lymphoblastic Leukaemia
Status: Recruiting | Type: Observational
Sponsor: Mats Heyman (Other)
Collaborators: Nordic Society for Pediatric Hematology and Oncology (Other); The Swedish Childhood Cancer Foundation (Unknown); NordForsk (Unknown)
Responsible Party: Sponsor-Investigator, Mats Heyman, MD, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: ALLTogether1 pilot
Record Dates: First submitted 2019-03-26; First posted 2019-04-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Acute Lymphoblastic
Keywords: Leukemia; Acute Lymphoblastic; ALL; ALLTogether; Leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood/blood plasma
  * Cerebrospinal fluid
  * Bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with newly diagnosed ALL
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational study - no intervention

SUMMARY:
The pilot study collects the experience of previously successful treatment of infants, children and young adults, with ALL from a number of well-renowned study groups into a new platform protocol, which is both a comprehensive system for stratification and treatment of ALL in this age-group as well as the basis for several randomised trials included in the study-design.

The pilot study is implemented as a master protocol without study specific interventions, thus as an observational study. The pilot study is for countries/study-groups who intend to join ALLTogether1 (including experimental interventions). For these countries the pilot study is crucial to optimise diagnostics, registration systems, collaborations with vendors, logistics and data-checks before starting the main study.

The study only includes "standard of care" treatment included in the master protocol.

DETAILED DESCRIPTION:
The aims of the ALLTogether study are to improve survival and quality of survival for children and young adults with ALL. ALL in young people has excellent outcome with >90% survival in children and about 75% in young adults. However, patients still die of disease - after relapse as a result of under-treatment.

Furthermore, a considerable fraction of younger patients are over-treated: All patients risk treatment-related death and some suffer long-term side-effects or secondary cancer. The rates of death from disease and death from therapy are almost the same for children. To show improvement with such good survival, large populations are needed.

Study groups from the five Nordic countries, Estonia and Lithuania (NOPHO), the UK (UKALL), the Netherlands (DCOG), Germany (COALL), Belgium (BSPHO), Ireland (PHOAI), Portugal (SHOP) and France (SFCE) have designed a common treatment protocol as new standard of care for children and young adults with ALL. The risk-stratification is based on a novel, personalised algorithm using clinical characteristics, genetic changes in the leukaemia and response to therapy.

The protocol will, based on a personalised risk-approach, define a platform for diagnosis and treatment onto which randomized as well as non-randomised interventions and translational studies can be added. This platform can also be used by countries joining the collaboration at a later date to prepare for full participation.

High-risk B-lineage patients may be stratified to Chimeric Antigen Receptor T-cell (CAR-T) therapy as an alternative to high-risk blocks and stem-cell transplant to reduce the side-effects.

Translational and other therapy-related research will be promoted by the common master protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with T-lymphoblastic (T-cell) or B-lymphoblastic precursor (BCP) leukaemia (ALL) according to the WHO-classification of Tumours of Haematopoietic and Lymphoid Tissues (Revised 4th edition 2017) and with a diagnosis confirmed by an accredited laboratory at a participating paediatric oncology or adult haematology centre.
* Age 0 - < 46 years (one day before 46th birthday) at the time of diagnosis, with the exception of infants with KMT2A-r BCP ALL (see exclusion criteria below).
* Patients with surface immunoglobulin negative (sIG-) BCP-ALL and an IG::MYC rearrangement, unless they have a concurrent BCL2/6 rearrangement. T-ALL patients with MYC translocations.
* Informed consent signed by the patient and/or parents/legal guardians according to country-specific age related guidelines
* The ALL diagnosis should be confirmed by an accredited laboratory at a participating paediatric oncology or adult haematology centre.
* The patient should be diagnosed and treated at a participating paediatric oncology or adult haematology centre in the participating countries.
* The patient should be a resident in one of the participating countries on a permanent basis or should intend to settle in a participating country, for instance by an application for asylum. Patients who are visiting the country as tourists should not be included. However, returning expatriots and patients who intend to stay at least for the duration of the treatment with primary diagnosis abroad may be included if no treatment has been administered and the diagnostic procedures are repeated at a participating centre.
* All women of childbearing potential (WOCBP) have to have a negative pregnancy test within 2 weeks prior to the start of treatment.

Exclusion Criteria:

* Age < 365 days and KMT2A-rearranged (KMT2A-r) BCP-ALL (documented presence of a KMT2A-split by FISH and/or a KMT2A fusion transcript). These patients will be transferred to an appropriate trial for infant KMT2A-r BCP-ALL, if available.
* Age >45 years at diagnosis.
* Patients with a previous malignant diagnosis (ALL as a second malignant neoplasm - SMN).
* Relapse of ALL.
* Patients with mature B-ALL (as defined by surface IG positivity) or any patients with IG::MYC and a concurrent BCL2/6 rearrangement.
* Patients with Ph-positive ALL (documented presence of t(9;22)(q34;q11) and/or of the BCR::ABL1 fusion transcript). These patients will be transferred to an appropriate trial for t(9;22) if available.
* Previously known ALL prone syndromes (e.g. Li-Fraumeni syndrome, germline ETV6 mutation), except for Down syndrome. Exploration for such ALL prone syndromes is not mandatory and patients in whom genetic work-up reveals a new germ-line mutation (index-cases) will remain in the study.
* Treatment with systemic corticosteroids corresponding to (>10mg prednisolone/m2/day) for more than one week and/or other chemotherapeutic agents in a 4-week interval prior to diagnosis (pre-treatment).
* Pre-existing contraindications to any treatment according to the ALLTogether protocol (constitutional or acquired disease prior to the diagnosis of ALL preventing adequate treatment).
* Any other disease or condition, as determined by the investigator, which could interfere with the participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with the study procedures.
* Women of childbearing potential who are pregnant at the time of diagnosis.
* Women of childbearing potential and fertile men who are sexually active and are unwilling to use adequate contraception during therapy. Efficient birth control is required, see section 18.9.
* Female patients, who are breast-feeding.
* Essential data missing from the registration of characteristics at diagnosis (in consultation with the protocol chair).

Ages: 0 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants 0-45 years with newly diagnosed acute lymphoblastic leukaemia. The protocol has no gender-bias. The total estimated recruitment in the pilot study is 500 participants.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) compared to historical controls | 5 year
Overall survival (OS) compared to historical controls | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Mats Heyman, M.D. PhD, Study Chair — Karolinska University Hospital
Locations (53):
- Denmark (6):
  - Aalborg University Hospital, Dept of Paediatrics, Aalborg
  - Aarhus University Hospital, Aarhus
  - Aarhus University Hospital, Child and Adolescent Health, Aarhus
  - Rigshospitalet, Dept of Haematology, Copenhagen
  - Rigshospitalet, Dept of Paediatrics, Copenhagen
  - Odense University Hospital, Dept of Paediatrics, Odense
- Estonia (3):
  - North Estonia Medical Centre, Dept of Haematology, Tallinn
  - Tallinn Children´s Hospital, Dept of Paediatrics, Tallinn
  - Tartu University Hospital, Tartu
- Finland (10):
  - Helsinki University Hospital, Dept of Haematology, Helsinki
  - Helsinki University Hospital, Dept of Paediatrics, Helsinki
  - Kuopio University Hospital, Dept of Haematology, Kuopio
  - Kuopio University Hospital, Dept of Paediatrics, Kuopio
  - Oulu University Hospital, Dept of Haematology, Dept of Medicine, Oulu
  - Oulu University Hospital, Dept of Paediatrics, Oulu
  - Tampere University Hospital, Dept of Haematology, Tampere
  - Tampere University Hospital, Dept of Paediatrics, Tampere
  - Turku University Hospital, Clinical Haematology and Stem Cell Transplantation Unit, Turku
  - Turku University Hospital, Dept of Paediatrics, Turku
- Landspitali University Hospital, Children's Hospital, Reykjavik, Iceland
- Lithuania (2):
  - Children's Hospital, Affiliate of Vilnius University Hospital, Vilnius
  - Vilnius University Hospital, Vilnius
- Norway (9):
  - Haukeland University Hospital, Dept of Haematology, Bergen
  - Haukeland University Hospital, Dept of Paediatrics, Bergen
  - Oslo University Hospital, Dept of Haematology, Oslo
  - Oslo University Hospital, Dept of paediatric haemato- and oncology, Oslo
  - Stavanger University Hospital, Dept of Haematology, Stavanger
  - University Hospital North Norway, Dept of Haematology, Tromsø
  - University Hospital of North Norway, Dept of Paediatrics, Tromsø
  - St. Olavs University Hospital, Dept of Paediatrics, Trondheim
  - St. Olavs University Hospital, Dept of Haematology, Trondheim
- Spain (9):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario San Joan de Déu, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Fuencarral-El Pardo
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Politécnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (13):
  - Sahlgrenska University Hospital, Section for Haematology and coagulation, Gothenburg
  - Sahlgrenska University Hospital, Dept of Paediatric Haematology and Oncology, Gothenburg
  - Linköping University Hospital, Dept of Haematology, Linköping
  - Linköping University Hospital, Dept of Paediatrics, Linköping
  - Skåne University Hospital, Dept of Haematology, Lund
  - Skåne University Hospital, Dept of Paediatrics, Lund
  - Örebro University Hospital, Section for Haematology, Örebro
  - Karolinska University Hospital, Dept of Paediatric Oncology and Haematology, Stockholm
  - Karolinska University Hospital, Patient area Haematology, Stockholm
  - Norrland University Hospital, Dept of Haematology, Umeå
  - Norrland University Hospital, Dept of Paediatrics, Umeå
  - Uppsala University Hospital, Dept of Haematology, Uppsala
  - Uppsala University Hospital, Dept of Paediatric Haematology and Oncology, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be entered into the study database. The data will be used to inform the coming main study regarding safety and overall outcomes of the master protocol. As such, these outcomes may be published in the context of a comparison with the ALLTogether1 protocol (the master protocol including experimental interventions, NCT 04307576, or compared with legacy protocols of the participating study-groups, The data of the pilot protocol will be shared according to the same principles as ALLTogether1 data.

REFERENCES:
- [Background] Toft N, Birgens H, Abrahamsson J, Griskevicius L, Hallbook H, Heyman M, Klausen TW, Jonsson OG, Palk K, Pruunsild K, Quist-Paulsen P, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Marquart HV, Madsen HO, Noren-Nystrom U, Schmiegelow K. Results of NOPHO ALL2008 treatment for patients aged 1-45 years with acute lymphoblastic leukemia. Leukemia. 2018 Mar;32(3):606-615. doi: 10.1038/leu.2017.265. Epub 2017 Aug 18. PMID 28819280
- [Background] Schramm F, Zimmermann M, Jorch N, Pekrun A, Borkhardt A, Imschweiler T, Christiansen H, Faber J, Feuchtinger T, Schmid I, Beron G, Horstmann MA, Escherich G. Daunorubicin during delayed intensification decreases the incidence of infectious complications - a randomized comparison in trial CoALL 08-09. Leuk Lymphoma. 2019 Jan;60(1):60-68. doi: 10.1080/10428194.2018.1473575. Epub 2018 Jul 3. PMID 29966458
- [Background] Mondelaers V, Suciu S, De Moerloose B, Ferster A, Mazingue F, Plat G, Yakouben K, Uyttebroeck A, Lutz P, Costa V, Sirvent N, Plouvier E, Munzer M, Poiree M, Minckes O, Millot F, Plantaz D, Maes P, Hoyoux C, Cave H, Rohrlich P, Bertrand Y, Benoit Y; Children-s Leukemia Group (CLG) of the European Organization for Research and Treatment of Cancer (EORTC). Prolonged versus standard native E. coli asparaginase therapy in childhood acute lymphoblastic leukemia and non-Hodgkin lymphoma: final results of the EORTC-CLG randomized phase III trial 58951. Haematologica. 2017 Oct;102(10):1727-1738. doi: 10.3324/haematol.2017.165845. Epub 2017 Jul 27. PMID 28751566
- [Background] Vora A, Goulden N, Wade R, Mitchell C, Hancock J, Hough R, Rowntree C, Richards S. Treatment reduction for children and young adults with low-risk acute lymphoblastic leukaemia defined by minimal residual disease (UKALL 2003): a randomised controlled trial. Lancet Oncol. 2013 Mar;14(3):199-209. doi: 10.1016/S1470-2045(12)70600-9. Epub 2013 Feb 7. PMID 23395119
- [Background] Pieters R, de Groot-Kruseman H, Van der Velden V, Fiocco M, van den Berg H, de Bont E, Egeler RM, Hoogerbrugge P, Kaspers G, Van der Schoot E, De Haas V, Van Dongen J. Successful Therapy Reduction and Intensification for Childhood Acute Lymphoblastic Leukemia Based on Minimal Residual Disease Monitoring: Study ALL10 From the Dutch Childhood Oncology Group. J Clin Oncol. 2016 Aug 1;34(22):2591-601. doi: 10.1200/JCO.2015.64.6364. Epub 2016 Jun 6. PMID 27269950
- [Derived] Fermer J, van Bunningen H, Zhou O, Abrahamsson J, Borssen M, Donner I, Heyman M, Holmqvist AS, Valind A, Vogt H, Ranta S, Harila A. Early Toxicity in Childhood Acute Lymphoblastic Leukemia: A Comparison of NOPHO ALL2008 and ALLTogether Protocols in Sweden. Pediatr Blood Cancer. 2025 Nov 20:e32168. doi: 10.1002/pbc.32168. Online ahead of print. PMID 41262029